CLINICAL TRIAL: NCT05736432
Title: Impacts of Wild Blueberries on Appetite and Weight Regulation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: San Diego State University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: HS-2023-001
Record Dates: First submitted 2023-02-09; First posted 2023-02-21 (Actual); Last update posted 2025-02-21 (Actual); Status verified 2025-02

CONDITIONS: Obesity; Weight Loss
Keywords: Blueberries; Yogurt; Weight loss; Appetite
MeSH Terms: conditions — Obesity; Weight Loss | interventions — blueberry extract

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Blueberries-Phase I (Experimental): feeding will consist of 1 C frozen wild blueberries along with ¾ C low-fat Mountain High yogurt (total energy intake=170 kcal)
  Interventions: Dietary Supplement: Blueberries
- Syrup-Phase I (Placebo Comparator): feeding will consist of an isocaloric feeding of ¾ C yogurt mixed with artificially flavored and colored blueberry syrup (Torani)
  Interventions: Dietary Supplement: Placebo
- Blueberries-Phase II (Experimental): 1 C frozen wild blueberries along with ¾ C low-fat Mountain High yogurt (total energy intake=170 kcal) along with a) dietary intervention, b) daily text messaging, and c) daily at-home weighing with a WiFi-enabled scale
  Interventions: Dietary Supplement: Blueberries
- Syrup-Phase II (Placebo Comparator): isocaloric feeding of ¾ C yogurt mixed with artificially flavored and colored blueberry syrup (Torani) along with a) dietary intervention, b) daily text messaging, and c) daily at-home weighing with a WiFi-enabled scale
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Blueberries — Experimental condition
  Arms: Blueberries-Phase I; Blueberries-Phase II
Dietary Supplement: Placebo — Placebo condition
  Arms: Syrup-Phase I; Syrup-Phase II

SUMMARY:
The objective is to complete a two-phase study to assess how wild blueberries impact regulation of appetite of overweight and obese men and women as well as to determine if wild blueberries can promote more effective weight loss than an isocaloric control. For phase I, the acute effects of consuming 1-cup of frozen wild blueberries mixed into ¾ C of low-fat yogurt will be compared to consuming an isocaloric serving of yogurt mixed with an artificially flavored and colored blueberry syrup. During acute testing, subjective ratings of appetite, glucose metabolism, and appetite-regulating hormones will be assessed. Phase II will consist of an 8-week feeding trial in which the same subjects will consume daily servings of yogurt mixed with either frozen wild blueberries or placebo syrup along with intensive counseling for weight loss. The hypothesis is that wild blueberries will reduce hunger by regulating appetite hormones and promoting beneficial glycemic and insulinemic responses and that daily consumption of wild blueberries will translate to improved adherence to a weight loss regimen and therefore greater weight and fat loss. Secondary aims for Phase II of this project will include exploring the impacts of blueberry consumption during weight loss on antioxidant status, inflammatory markers, blood lipid profiles, glucose status, dietary intake, physical activity and blood pressure.

DETAILED DESCRIPTION:
For Phase I, all subjects will complete two acute feeding trials in random order. One feeding will consist of 1 C frozen wild blueberries along with ¾ C low-fat Mountain High yogurt (total energy intake=170 kcal). The other feeding will consist of an isocaloric feeding of ¾ C yogurt mixed with artificially flavored and colored blueberry syrup (Torani). A standardized meal will be consumed the evening prior to testing to minimize fluctuations during the testing days. Arterialized fingerprick blood samples from heated hands will be collected into Greiner Bio-One MiniCollect™ Capillary Blood Collection System Tubes containing Ethylenediaminetetraacetic acid while fasted and 30, 60 and 120 minutes after food intake for analysis of glucose, insulin, ghrelin, and pancreatic peptide. Appetitive responses (hunger, fullness, desire to eat, and prospective food consumption) will be assessed by 100-mm visual analog scales at baseline and 15, 30, 45, 60, 90, and 120 minutes after intake.

For Phase II, subjects will be equally divided and matched for body fatness into two randomly assigned groups. Both groups will be counseled for weight loss, which will be achieved through a comprehensive program including a) dietary intervention, b) daily text messaging, and c) daily at-home weighing with a WiFi-enabled scale. In addition, groups will be randomly assigned to daily consume the same 170 kcal yogurt parfait described above containing either wild blueberries or placebo as an afternoon snack for 8 weeks. The rationale for the inclusion of a healthy, wild blueberry in yogurt afternoon snack intervention is supported by the National Health And Nutrition Examination Survey analyses that revealed a shift in eating patterns towards the evening in combination with an increase in snacking occasions, particularly in the afternoon/evening hours. Further, the majority of the snacking occasions include unhealthy, high fat/high sugar foods, potentially contributing to unwanted weight gain and obesity. Moreover, since blueberries can elevate pancreatic peptide for at least 2 hours after consumption, this could enhance the likelihood of maintaining lower intake during the evening meal. Thus, overall, it is proposed that the afternoon wild blueberry/yogurt snack will promote satiety and reduce overeating (especially of unhealthy foods) later in the day.

All participants will be counseled to achieve a 500-kcal/d energy deficit (from their baseline eucaloric diet). Energy requirements will be estimated by calculating resting metabolic rate using the equations of Schofield and multiplying by an activity factor of 1.3. The participants will meet with investigators every two-weeks for intensive counseling to ensure adherence to the dietary prescription. Before and after the trial, fasted blood will be collected into tubes for both plasma and serum to assess total antioxidant capacity, C-reactive protein, blood lipid concentrations, glucose and insulin. During lab visits investigators will assess anthropometrics (height, body weight, and body composition via dual x-ray absorptiometry, dietary intake, physical activity behaviors, food cravings, and blood pressure. Adequate samples of blood will be collected to allow us to bank plasma for future analyses if additional funding is obtained in the future.

ELIGIBILITY:
Inclusion Criteria:

* Overweight or Obese (BMI 25-40)

Exclusion Criteria:

* Pregnancy
* Smoking
* >5 kg wt fluctuation in the past 3 months
* exercising > 2 times per week
* Medical conditions or medications that may affect body weight, metabolism, other outcome measures
* Allergy to blueberries or yogurt
* Already eating blueberries more than twice weekly
* Consumption of >50 g/d alcohol

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2023-03-01 (Actual); Primary Completion 2024-11-01 (Actual); Study Completion 2025-02-01 (Actual)

PRIMARY OUTCOMES:
Plasma Glucose | 8 weeks
  fasted
Total Cholesterol | 8 weeks
  Total Cholesterol
Triglycerides | 8 weeks
  Triglycerides
HDL-Cholesterol | 8 weeks
  HDL-Cholesterol
Insulin | 8 weeks
  Insulin
Ghrelin | 8 weeks
  Ghrelin
Pancreatic peptide | 8 weeks
  Pancreatic peptide
C-Reactive Protein | 8 weeks
  C-Reactive Protein
Total Antioxidant Capacity | 8 weeks
  Colorimetric assay kit using blood serum
Blood Pressure | 8 weeks
  Systolic and Diastolic
Body Composition | 8 weeks
  Daily via bioimpedance Wifi Scales
Body Composition | 8 weeks
  dual x-ray absorptiometry

CONTACTS AND LOCATIONS:
Overall Officials: Shirin Hooshmand, PhD, RD, Study Director — San Diego State University
Locations (1):
- Mark Kern, PhD, RD, San Diego, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Stote K, Corkum A, Sweeney M, Shakerley N, Kean T, Gottschall-Pass K. Postprandial Effects of Blueberry (Vaccinium angustifolium) Consumption on Glucose Metabolism, Gastrointestinal Hormone Response, and Perceived Appetite in Healthy Adults: A Randomized, Placebo-Controlled Crossover Trial. Nutrients. 2019 Jan 19;11(1):202. doi: 10.3390/nu11010202. PMID 30669469
- [Background] Molan AL, Lila MA, Mawson J. Satiety in rats following blueberry extract consumption induced by appetite-suppressing mechanisms unrelated to in vitro or in vivo antioxidant capacity. Food Chemistry. 2008 Apr 1;107(3):1039-44.
- [Background] James LJ, Funnell MP, Milner S. An afternoon snack of berries reduces subsequent energy intake compared to an isoenergetic confectionary snack. Appetite. 2015 Dec;95:132-7. doi: 10.1016/j.appet.2015.07.005. Epub 2015 Jul 7. PMID 26162950
- [Background] DeFuria J, Bennett G, Strissel KJ, Perfield JW 2nd, Milbury PE, Greenberg AS, Obin MS. Dietary blueberry attenuates whole-body insulin resistance in high fat-fed mice by reducing adipocyte death and its inflammatory sequelae. J Nutr. 2009 Aug;139(8):1510-6. doi: 10.3945/jn.109.105155. Epub 2009 Jun 10. PMID 19515743
- [Background] Elks CM, Terrebonne JD, Ingram DK, Stephens JM. Blueberries improve glucose tolerance without altering body composition in obese postmenopausal mice. Obesity (Silver Spring). 2015 Mar;23(3):573-80. doi: 10.1002/oby.20926. Epub 2015 Jan 22. PMID 25611327
- [Background] Nair AR, Elks CM, Vila J, Del Piero F, Paulsen DB, Francis J. A blueberry-enriched diet improves renal function and reduces oxidative stress in metabolic syndrome animals: potential mechanism of TLR4-MAPK signaling pathway. PLoS One. 2014 Nov 5;9(11):e111976. doi: 10.1371/journal.pone.0111976. eCollection 2014. PMID 25372283
- [Background] Roopchand DE, Kuhn P, Rojo LE, Lila MA, Raskin I. Blueberry polyphenol-enriched soybean flour reduces hyperglycemia, body weight gain and serum cholesterol in mice. Pharmacol Res. 2013 Feb;68(1):59-67. doi: 10.1016/j.phrs.2012.11.008. Epub 2012 Dec 4. PMID 23220243
- [Background] Seymour EM, Tanone II, Urcuyo-Llanes DE, Lewis SK, Kirakosyan A, Kondoleon MG, Kaufman PB, Bolling SF. Blueberry intake alters skeletal muscle and adipose tissue peroxisome proliferator-activated receptor activity and reduces insulin resistance in obese rats. J Med Food. 2011 Dec;14(12):1511-8. doi: 10.1089/jmf.2010.0292. Epub 2011 Aug 23. PMID 21861718